CLINICAL TRIAL: NCT00020995
Title: Effects of a Low Fat Diet on Serum Factors and Prostate Cancer
Brief Title: Low-Fat, High-Fiber Diet Compared to a Standard Diet in Treating Patients With Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Prevention
Other Study IDs: CDR0000068737; UCLA-0001030; NCI-G01-1973
Record Dates: First submitted 2001-07-11; First posted 2003-01-27 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2004-05

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage I prostate cancer; stage IIB prostate cancer; stage IIA prostate cancer; stage III prostate cancer; stage IV prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

INTERVENTIONS:
Procedure: therapeutic dietary intervention

SUMMARY:
RATIONALE: A low-fat, high-fiber diet may slow the growth of prostate cancer.

PURPOSE: Randomized phase II trial to compare the effectiveness of a low-fat, high-fiber diet with that of a standard diet in treating patients who have prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the inhibition of growth of human prostate cancer cell lines by serum from patients with prostate cancer before and after being fed a low fat, high fiber diet.
* Determine the underlying mechanism through which a low fat, high fiber diet affects the growth of prostate cancer cell lines.
* Determine whether a low fat, high fiber diet inhibits the growth of prostate cancer cell lines through androgen-dependent and/or androgen- independent mechanisms in these patients.
* Determine the growth factors, hormones, and/or binding proteins that may be responsible for affecting the growth of prostate cancer cell lines in these patients.

OUTLINE: This is a randomized study. Patients are randomized to 1 of 2 arms.

* Arm I: Patients receive a low fat, high fiber diet daily for 3 weeks.
* Arm II: Patients receive a control diet containing the standard amounts of fat and fiber.

PROJECTED ACCRUAL: A total of 40 patients (20 per arm) will be accrued for this study within 6 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of adenocarcinoma of the prostate
* Previously untreated and on watchful waiting
* Medically able to receive dietary intervention

PATIENT CHARACTERISTICS:

Age:

* 40 to 80

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* Must be willing to travel to UCLA 3 days a week for 4 weeks to obtain specially prepared foods

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Not specified

Endocrine therapy:

* No concurrent luteinizing hormone-releasing hormone agonists (leuprolide or goserelin)
* No concurrent androgen-receptor blocking agents (flutamide or bicalutamide)
* No concurrent testosterone
* No concurrent insulin
* No concurrent finasteride

Radiotherapy:

* Not specified

Surgery:

* No prior orchiectomy

Other:

* No concurrent saw palmetto supplement

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-08; Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Aronson, MD, Study Chair — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California, United States

REFERENCES:
- [Result] Aronson WJ, Barnard RJ, Freedland SJ, Henning S, Elashoff D, Jardack PM, Cohen P, Heber D, Kobayashi N. Growth inhibitory effect of low fat diet on prostate cancer cells: results of a prospective, randomized dietary intervention trial in men with prostate cancer. J Urol. 2010 Jan;183(1):345-50. doi: 10.1016/j.juro.2009.08.104. PMID 19914662